CLINICAL TRIAL: NCT02397564
Title: Treatment of Post-Surgical Scars With Traditional Ablative Er:YAG Versus Fractional Ablative Er:YAG
Acronym: Er:YAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14.1075
Record Dates: First submitted 2015-03-04; First posted 2015-03-25 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Post-Surgical Scars
Keywords: scar; ICD-10 CM:L90.5
MeSH Terms: conditions — Cicatrix | interventions — Lasers, Solid-State

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Enroll 20 patients for nonsurgical treatment of surgical scars. Half of each scar will be treated with the Er:YAG laser on the traditional ablative setting and the other half of the scar will receive Er:YAG treatment with the fractional ablative setting. The patients will receive 3 treatments at monthly intervals. They will follow up at 1 and 2 months after the treatment.
  Interventions: Device: Er:YAG laser, traditional and fractional settings

INTERVENTIONS:
Device: Er:YAG laser, traditional and fractional settings — Half the scar will be treated with traditional ablative setting and the other half will be treated with the fractional ablative setting

SUMMARY:
The investigators will compare the efficacy of Traditional Ablative Er:YAG Versus Fractional Ablative Er:YAG in a split scar study. The patient will receive a month treatment for 3 months. Then follow up for the next 2 months.

DETAILED DESCRIPTION:
Background: Scars are a common complaint of patients at presentation to a dermatology office. To optimize cosmetic results, the investigators propose to compare erbium-doped yttrium aluminium garnet (Er:YAG) laser therapy on two different settings: traditional ablative versus fractional ablative. A side to side comparison of split scars will be done to evaluate the two settings. Fractionated photothermolysis (fractional setting) has improved the field of laser surgery by allowing the surgery to target microscopic treatment zones (MTZ). MTZ's allow for cylinders of damage created by laser surgery to be surrounded by normal, unaffected skin. This acts as a reservoir for healing and allows for the microwounds created by laser treatment to heal quickly and with minimal discomfort.

Objective: To compare efficacy and cosmetic appearance of scars treated with Er:YAG ablative laser on traditional ablative resurfacing setting versus fractional ablative resurfacing setting.

Methods: Enroll 20 patients for nonsurgical treatment of surgical scars. Half of each scar will be treated with the Er:YAG laser on the traditional ablative setting and the other half of the scar will receive Er:YAG treatment with the fractional ablative setting. The patients will receive 3 treatments at monthly intervals. They will follow up at 1 and 2 months after the treatment. Pictures of the scar will be taken at a 45 degree and 90 degree angle at baseline, before each treatment, after each treatment, and at all follow up appointments. The patients will be blinded as to which side is treated with which laser setting. At the end of the trial, they will be offered the chance to have the side they felt had less improvement treated with the laser device that had been used on the contralateral side of the scar.

Results: A panel of three blinded dermatologists will evaluate the scar on a well-established five point grading scale for erythema, height and texture, and overall cosmetic outcome. The mean, standard deviation, and kappa values will be calculated. Patients will be asked the same scar evaluation questions as the panel as well as their overall satisfaction, how much pain was associated with the procedure, which laser they preferred, and would they recommend treatment to a friend or family member.

ELIGIBILITY:
Inclusion Criteria:

* over 8 weeks s/p scar
* linear closure
* visibly symmetric scar
* over 18 years old

Exclusion Criteria:

* concomitant treatment of involved skin
* propensity for keloid scarring
* use of oral retinoids for the past 1 year
* pregnancy
* immunosuppression
* prior laser to the area

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy S Brown, MD, Principal Investigator — University of Louisville

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group: Enroll 20 patients for nonsurgical treatment of surgical scars. Half of each scar will be treated with the Er:YAG laser on the traditional ablative setting and the other half of the scar will receive Er:YAG treatment with the fractional ablative setting. The patients will receive 3 treatments at monthly intervals. They will follow up at 1 and 2 months after the treatment.
  Er:YAG laser, traditional and fractional settings: Half the scar will be treated with traditional ablative setting and the other half will be treated with the fractional ablative setting
Period: Overall Study
Arm/Group | Intervention Group
Started | 20
Completed | 16
Not Completed | 4

BASELINE CHARACTERISTICS:
Groups:
- Treatment Group: Enroll 20 patients for nonsurgical treatment of surgical scars. Half of each scar will be treated with the Er:YAG laser on the traditional ablative setting and the other half of the scar will receive Er:YAG treatment with the fractional ablative setting. The patients will receive 3 treatments at monthly intervals. They will follow up at 1 and 2 months after the treatment.
  Er:YAG laser, traditional and fractional settings: Half the scar will be treated with traditional ablative setting and the other half will be treated with the fractional ablative setting
Arm/Group | Treatment Group
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 46 [28 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Region of Enrollment [Number; unit: participants] — Patients enrolled in a consecutive order from our surgical log book.
  participants
    United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Patient Observer Scar Assessment Scale (POSAS)
Description: It uses a 10-point scoring system with a score of 1 representing a normal-appearing skin and a score of 10 representing the worst possible scar. Total scores range from 6 to 60 with the lower score indicate a better outcome.
Time Frame: 5 months
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Treatment Group: Subjects receiving treatment for scar
Arm/Group | Treatment Group
Number analyzed (Participants) | 16
units on a scale
  Physician Fully Ablative Laser | 17.69 (2.03)
  Physician Fractionated Laser | 11.2 (2.03)
  Patients Fully Ablative Laser | 15.2 (1.58)
  Patients Fractionated Laser | 11.4 (1.58)
Statistical Analysis 1: Comparison: Treatment Group; Test type: Superiority or Other; p = 0.019, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Patient Preference
Description: The number of patients who preferred the fractionated laser
Time Frame: 5 months
Population: Those who expressed a preference.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Group: Number of patients that preferred the fractionated laser.
Arm/Group | Treatment Group
Number analyzed (Participants) | 16
Participants | 15

ADVERSE EVENTS:
Time Frame: 5 months
Groups:
- Treatment Group: Those who went laser treatment.
Arm/Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No